CLINICAL TRIAL: NCT02374671
Title: A Prospective, Multicenter Clinical Trial of the VisAbility Micro Insert System for Improvement of Near Visual Acuity In Presbyopic Patients
Brief Title: A Clinical Trial of The VisAbility Micro Insert System for Presbyopic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Refocus Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VIS-2014
Record Dates: First submitted 2015-02-17; First posted 2015-03-02 (Estimated); Results first posted 2020-01-06 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2019-12

CONDITIONS: Presbyopia
Keywords: Near Vision; Reading Vision; Reading Glasses; Reading; Readers; Presbyopic; Presbyopia
MeSH Terms: conditions — Presbyopia; Myopia

STUDY DESIGN:
Intervention Model Description: A non-randomized arm was run in parallel with a randomized sub-study consisting of 2 arms; Immediate Treatment and Deferred Treatment. Upon completion of the 6 month observation period, the Deferred Treatment group then crosses over upon implantation to become part of the overall study group.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Implantation-Non-Randomized (Experimental): Subjects are not participants in the randomized sub-study. VisAbility micro inserts surgically implanted in the eye(s) after enrollment and meeting inclusion/exclusion criteria.
  Interventions: Device: VisAbility Micro Insert
- Implantation-Randomized (Experimental): Subjects are participants in the randomized sub-study. Subjects were randomized to the Immediate Treatment group. VisAbility micro inserts surgically implanted in the eyes. Subjects are participants in the randomized sub-study after enrollment and meeting inclusion/exclusion criteria.
  Interventions: Device: VisAbility Micro Insert
- Deferred Implantation-Randomized (No Intervention): Subjects are participants in the randomized sub-study after enrollment and meeting inclusion/exclusion criteria. Subjects were randomized to the Deferred Treatment group are observed for 6 months. Upon completion of the observation follow-up, subjects can opt to have VisAbility micro inserts surgically implanted in the eye(s) and become part of the overall study experimental group.

INTERVENTIONS:
Device: VisAbility Micro Insert — Subjects are implanted with the VisAbility Micro Insert (Model SGP-046) and followed for 24 months.
  Arms: Implantation-Non-Randomized; Implantation-Randomized

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the VisAbility Micro Insert System for the improvement of near visual acuity in presbyopic patients.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the safety and effectiveness of the VisAbility Implant System (VIS) for the improvement of near visual acuity in presbyopic patients. This is a prospective clinical study that enrolled a total of 360 subjects ranging in age between 45 and 60 years of age at 13 clinical sites. Subjects were implanted with the VisAbility Implant model SGP-046 in the primary eye and then in the fellow eye no sooner than 14 days later. Subjects were examined at one day, one week and at 1, 2, 3, 6, 12, 18 and 24 months post-operatively.

The study also included a 60 subject randomized controlled sub-study at 3 investigation sites. Sub-study subjects were randomized (1:1 ratio) to a surgery group or a control group. Subjects randomized to the surgery group underwent surgery and were followed for 24 months in the same manner as the larger non-randomized surgical group. Subjects randomized to the control group were observed for 6 months, and were then eligible to undergo surgery after completion of this 6-month observation period.

The primary endpoint is the achievement of distance corrected near visual acuity (DCNVA) of Snellen equivalent 20/40 or better (at 40 cm) and at least 10 letters (ETDRS) improvement in DCNVA in the primary eye.

This endpoint is evaluated against two objectives, a) 75% or more of primary eyes achieve the effectiveness endpoint at 12 months postoperative and b) the percentage of primary eyes achieving the effectiveness endpoint at 6 months postoperative (6-month responder rate) is higher than the percentage in the randomized control group.

Safety data analyses were performed and separate summaries are provided for primary and all eyes. Descriptive statistics on the following attributes are provided for; BCDVA, IOP, Slit lamp findings, Fundus exam findings, and Adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a Best Corrected Distance Visual Acuity (BCDVA) of 20/20 in each eye
* Subjects must have a Distance Corrected Near Visual Acuity (DCNVA) @ 40 cm of 20/50, 20/63, or 20/80 in each eye
* Subjects must have an Uncorrected Near Visual Acuity (UCNVA) @ 40 cm of 20/50, 20/63, or 20/80 in each eye
* Subject's Preoperative Manifest Refraction Spherical Equivalent (MRSE) in each eye must be -0.75 to +0.50 diopters with no more than 1.00 diopter of astigmatism.
* Cycloplegic refraction spherical equivalent (CRSE) difference from MRSE should be less than or equal to 0.50 diopters.
* Subjects must require a minimum add of +1.25 or greater to read 20/20 at near (40 cm).
* Subjects must be alert, mentally competent, and able to understand and comply with the requirements of the clinical study, and be personally motivated to abide by the requirements and restrictions of the clinical study. Patients must be available for the follow-up period.
* Subjects must be able to provide written informed consent

Exclusion Criteria:

* Pupil has a baseline percent change from scotopic to photopic of less than 30% or an absolute difference of less than 1.00 mm between scotopic and photopic pupil size as measured by the NeurOptics Pupillometer
* Subjects with ocular inflammation, chronic uveitis, or other recurrent anterior or posterior segment inflammatory conditions in either eye; subjects with any ocular or systemic disease(s) posing a significant risk for ocular inflammation including but not limited to, autoimmune disorders (e.g. rheumatoid arthritis, ankylosing spondylitis, Reiter's syndrome, ulcerative colitis, Chron's disease, psoriasis, sarcoidosis, Bechet's disease), infections (toxoplasmosis, cat-scratch fever, West Nile virus, syphilis, tuberculosis, herpes zoster, herpes simplex, adenovirus), ocular trauma or gout.
* Subjects with scleral thickness of less than 530 microns as measured 3.5 to 40.00 mm posterior to the superior temporal quadrant limbus in either eye.
* Subjects with a history of any prior intraocular procedure (e.g. corneal transplant, filtering procedures for glaucoma, vitrectomy, retinal detachment repair, cataract surgery) or any prior refractive procedure (e.g. LASIK (laser in situ keratomileusis), surface excimer, or incisional surgery) in either eye.
* Subjects with any history of prior extraocular muscle surgery or orbital surgery.
* Subjects with chronic ocular disease including but not limited to corneal pathology, primary or secondary glaucoma, iritis, herpes simplex, uveitis, trachoma, ocular pemphigoid, Sjogrens disease, uveal melanoma, Thyroid Related Immune Orbitopathy or clinical significant retinal pathology in either eye.
* Subjects with any acute ocular disease that has not been completely treated and resolved for at least three months such as conjunctivitis, blepharitis, chalazion, corneal abrasion or keratitis in either eye.
* Subjects with chronic systemic diseases which may affect the eye, including but not limited to diabetes, ulcerative colitis, systemic lupus erythematosus, Chron's disease, collagen vascular disease, rheumatoid arthritis, any bleeding diathesis, or systemic manifestations of HIV/AIDS. Any other uncontrolled systemic disease (e.g. hypertension, cancer, etc.) that could compromise the patient's participation.
* Use of any medication such as Coumadin, that could make the surgical procedure more difficult. Subjects using Coumadin, aspirin, or NSAID (non-steroidal anti inflammatory drug) medications under orders from a doctor must be able to provide written approval from the treating doctor for discontinuing this medication at least 10 days prior to surgery.
* Subjects with chronic ocular surface disease, including but not limited to subjects with a prior diagnosis of chronic dry eye syndrome based on tests such as but not limited to, corneal or conjunctival staining, Ocular surface Disease Index symptom score or Schirmer tear testing.
* Subjects who are allergic to any medications used in the protocol
* Subjects who are pregnant, lactating, or of child-bearing age adn not practicing a medically approved method of birth control.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 365 (Actual)
Dates: Start 2014-11-15 (Actual); Primary Completion 2018-04-13 (Actual); Study Completion 2018-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Selene Burke, O.D., Study Director — V.P. Clinical Affairs
Locations (14):
- United States (14):
  - Coastal Vision, Orange, California
  - Gordon Weiss Vision Institute, San Diego, California
  - Aloha Laser Vision, Honolulu, Hawaii
  - The Midwest Center for Sight, Des Plaines, Illinois
  - Eye Surgeons Of Indiana PC, Indianapolis, Indiana
  - Eye Care Institute, Louisville, Kentucky
  - Chu Vision Institute, Bloomington, Minnesota
  - South Shore Eye Care LLP, Wantagh, New York
  - South Shore Eye Care, LLP, Wantagh, New York
  - Physicians Protocol, Greensboro, North Carolina
  - Comprehensive EyeCare of Central Ohio, Westerville, Ohio
  - Bucci Laser Vision, Wilkes-Barre, Pennsylvania
  - Key Whitman Eye Center, Dallas, Texas
  - Braverman-Terry-Oei Eye Associates, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor Website — http://www.refocus-group.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The prospective, multicenter clinical trial of the VisAbility micro insert was conducted at 13 clinical sites. All recruitment evaluations were performed at the Principal Investigator's sites and subjects were screened for eligibility. If inclusion/exclusion criteria were met, informed consent was obtained and the subject was enrolled in the study.
Pre-assignment Details: Once determined eligible and informed consent was obtained, both eyes were enrolled in the study. Per protocol, primary outcome analysis must be performed on the primary eye only and the primary eye is therefore the unit of analysis. Fellow eyes were followed for safety outcomes and summarized separately.
Units Other Than Participants: Eye
Groups:
- Implantation-Non-Randomzied: Subjects are not participants in the randomized sub-study. VisAbility micro inserts surgically implanted in the eye(s) after enrollment and meeting inclusion/exclusion criteria.
  VisAbility Micro Insert: Subjects are implanted with the VisAbility Micro Insert (Model SGP-046) and followed for 24 months.
- Deferred Implantion-Randomized: Subjects are participants in the randomized sub-study after enrollment and meeting inclusion/exclusion criteria. Subjects were randomized to the Deferred Treatment group are observed for 6 months. Upon completion of the observation follow-up, subjects can opt to have VisAbility micro inserts surgically implanted in the eye(s) and become part of the overall study experimental group.
Period: Observation (Deferred Implantation)
Arm/Group | Implantation-Non-Randomzied | Implantation-Randomized | Deferred Implantion-Randomized
Started | 0; 0 Eye | 0; 0 Eye | 31; 62 Eye
Completed | 0; 0 Eye | 0; 0 Eye | 26; 52 Eye
Not Completed | 0; 0 Eye | 0; 0 Eye | 5; 10 Eye
Not completed — Withdrawal by Subject | 0 | 0 | 4
Not completed — Adverse Event | 0 | 0 | 1
Period: Implantation- Nonrandomized & Randomized
Arm/Group | Implantation-Non-Randomzied | Implantation-Randomized | Deferred Implantion-Randomized
Started | 306; 604 Eye ((8) subjects were unilaterally implanted) | 28; 55 Eye ((1) subject was unilaterally implanted) | 26; 49 Eye ((3) subjects were unilaterally implanted)
Completed | 281; 571 Eye | 27; 53 Eye | 23; 44 Eye ((1) unilaterally implanted subject discontinued (1 eye))
Not Completed | 25; 33 Eye | 1; 2 Eye | 3; 5 Eye
Not completed — Lost to Follow-up | 17 | 1 | 2
Not completed — Adverse Event | 7 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Implantation-Non-Randomized | Implantation-Randomized | Deferred Implantion-Randomized | Total
Number analyzed (Participants) | 306 | 28 | 26 | 360
Age, Continuous [Mean (Full Range); unit: years] | 51.8 [45 to 60] | 50.1 [45 to 58] | 51.0 [45 to 58] | 51.6 [45 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 10 | 9 | 143
  Male | 182 | 18 | 17 | 217
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 9 | 9 | 38
  Not Hispanic or Latino | 283 | 19 | 17 | 319
  Unknown or Not Reported | 3 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 17 | 1 | 0 | 18
  Native Hawaiian or Other Pacific Islander | 4 | 0 | 0 | 4
  Black or African American | 14 | 0 | 1 | 15
  White | 262 | 23 | 22 | 307
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 9 | 4 | 3 | 16
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 306 | 28 | 26 | 360
DCNVA 20/40 or Better (at baseline) [Count of Participants; unit: Participants] | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Primary Eyes With Distance Corrected Near Visual Acuity (DCNVA) to 20/40 or Better and Gain of At Least 10 Letters.
Description: Measurement of the Distance Corrected Near Visual Acuity at 40 centimeters achieving 20/40 or better and Gain of At Least 10 Letters at 24 months for the primary eye.
Time Frame: From date of baseline measurement until the date of study withdrawal or study completion, whichever came first, assessed up to 2 years.
Population: Explanted primary eyes were analyzed as failures. Data for primary eyes that missed the 24 month visit, were lost to follow-up, or withdrew consent prior to the 24 month visit were not imputed. Per protocol, primary outcome analysis must be performed on the primary eye only. Fellow eye data is used for safety outcomes and summarized separately.
Measure: Count of Participants; unit: Participants
Groups:
- Overall Study Population: A total of 360 subjects at 14 sites received implantation of VisiAbility micro inserts and were followed for 24 months post surgical. As per the protocol, the primary eye is the unit of analysis and was used for primary endpoint analysis. Fellow eyes were followed for safety and summarized separately. The primary eyes of subjects participating in the randomized sub-study were analyzed separately, though, they were also considered part of the overall study if they received implantation of the micro inserts.
Arm/Group | Overall Study Population
Number analyzed (Participants) | 344
Participants | 289

2. Secondary Outcome: Number of Primary Eyes With DCNVA 20/40 of Better and Gain of 10 Letters More at 6 Months for the Randomized Substudy
Description: The randomized surgery group is defined as successful if the percentage of primary eyes achieving Distance Corrected Near Visual Acuity at 40 centimeters of 20/40 of Better and Gain of 10 Letters more at 6 months postoperative (i.e. 6-month responder rate) is higher than the percentage in the randomized control group.
Time Frame: From date of randomization until the date of study withdrawal or sub-study completion at 6 months, whichever came first.
Measure: Count of Participants; unit: Participants
Arm/Group | Implantation-Randomized | Deferred Implantion-Randomized
Number analyzed (Participants) | 28 | 29
Participants | 18 | 2

ADVERSE EVENTS:
Time Frame: Adverse event reporting continued through 24 months.
Description: An Adverse Event ("AE") is any untoward sign, symptom or disease observed during the course of the study regardless of the suspected cause. Conditions or diseases that are pre-existing or chronic but stable are not Adverse Events. Changes in pre-existing or chronic conditions or diseases that are consistent with natural disease progression are not Adverse Events.
Groups:
- VisAbility Micro Insert Implantation - Single Arm: For post-implant safety analysis, the Implantation-Non Randomized, Implantation-Randomized, and Deferred Implantation-Randomized arms were combined into (one) safety cohort (306 subjects + 26 subjects + 28 subjects, respectively), per protocol. All 360 implanted subjects that received the VisAbility Micro Insert implantation were followed for 24 months and were not analyzed separately. I.e. Subjects who participated in the randomized sub-study crossed over into a single (safety) arm at the time of implantation. For safety analysis and adverse event reporting, all implanted subjects were considered one cohort as there was no difference in treatment nor follow-up after VisAbility Micro Insert implantation.
Arm/Group | VisAbility Micro Insert Implantation - Single Arm
All-Cause Mortality (participants affected / at risk) | 0/360
Serious Adverse Events (participants affected / at risk) | 4/360
Other Adverse Events (participants affected / at risk) | 170/360
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VisAbility Micro Insert Implantation - Single Arm (N=360)
Serious Ocular Adverse Events (Eye disorders) | 0 (0) — Any Serious Ocular Adverse Events
Serious Non-Ocular Adverse Events (General disorders) | 4 (4) — Any Serious Non-Ocular Adverse Events
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VisAbility Micro Insert Implantation - Single Arm (N=360)
Visual Acuity (Eye disorders) | 9 (10)
Lid (Eye disorders) | 33 (64)
Cornea/Conjunctiva (Eye disorders) | 89 (159)
Iris/Pupil (Eye disorders) | 1 (1)
Anterior Chamber (Eye disorders) | 8 (9)
Lens (Eye disorders) | 2 (3)
Sclera (Intraoperative Events) (Eye disorders) | 8 (8)
Intraocular Pressure (Eye disorders) | 6 (6)
Fundus/Posterior Pole (Eye disorders) | 3 (3)
Secondary Surgical Intervention (Surgical and medical procedures) | 23 (28)
Allergic Reactions to Medications (Surgical and medical procedures) | 2 (4)
Other (Eye disorders) | 50 (70)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study.

The Sponsor encourages publication and presentation of the safety and effectiveness results upon completion of the study. Per the established agreement, the Principal Investigators will work with the Sponsor, in good faith, to ensure all confidential and proprietary information is redacted.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-03): https://cdn.clinicaltrials.gov/large-docs/71/NCT02374671/Prot_SAP_000.pdf